CLINICAL TRIAL: NCT03046498
Title: Addressing Diabetes Together: Implementation of a Regional Partnership for Population Health Management in Southeast Minnesota
Brief Title: Addressing Diabetes Together
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Aaron L. Leppin, M.D., WellConnect Medical Director, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-008948
Record Dates: First submitted 2017-02-02; First posted 2017-02-08 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Program participants (Experimental): Patients enrolled in the DSMP and DPP who provide consent.
  Interventions: Behavioral: Evidence-Based Program

INTERVENTIONS:
Behavioral: Evidence-Based Program — DSMP and DPP

SUMMARY:
Integration of Diabetes Prevention Program (DPP) and Diabetes Self Management Program (DSMP) into WellConnect.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* Diagnosis of diabetes
* enrolled in the DSMP or DPP

Exclusion Criteria:

* unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Measure change in number of program offerings implemented in the community | Change from Baseline to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Leppin AL, Okamoto JM, Organick PW, Thota AD, Barrera-Flores FJ, Wieland ML, McCoy RG, Bonacci RP, Montori VM. Applying Social Network Analysis to Evaluate Implementation of a Multisector Population Health Collaborative That Uses a Bridging Hub Organization. Front Public Health. 2018 Nov 2;6:315. doi: 10.3389/fpubh.2018.00315. eCollection 2018. PMID 30450355